CLINICAL TRIAL: NCT01082861
Title: A Phase 4, Randomized, Open Label Clinical Trial to Determine Efficacy and Immunomodulation of Simultaneous HPV/HBV Vaccination Tango-trial)
Brief Title: Efficacy and Immunomodulation Study of Simultaneous Human Papillomavirus/ Hepatitis B (HPV/HBV) Vaccination
Acronym: TANGO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to recent strategic policy developments in the national vaccination program it is uncertain preadolescent girls will receive the HBV vaccin.
Sponsor: National Institute for Public Health and the Environment (RIVM) (Other Government)
Responsible Party: Hein Boot, section head LIS, Institute of Public Health and the Environment
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LIS144; 2010-018459-86 (EudraCT Number)
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2010-03

CONDITIONS: Human Papillomavirus Infection
Keywords: 1998 female birth cohort eligible for HPV vaccination in 2011 within the Dutch NIP
MeSH Terms: conditions — Papillomavirus Infections | interventions — human papillomavirus vaccine, L1 type 16, 18; Engerix-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- HPV&HBV vaccin (Experimental): HPV&HBV vaccin
  Interventions: Biological: Cervarix; Biological: Engerix-B
- HPV vaccination (Experimental): HPV vaccination
  Interventions: Biological: Cervarix
- HBV vaccination (Experimental): HBV vaccination
  Interventions: Biological: Engerix-B

INTERVENTIONS:
Biological: Cervarix — Cervarix, HPV vaccin
  Arms: HPV vaccination; HPV&HBV vaccin
Biological: Engerix-B — Engerix-B, HBV vaccin
  Arms: HBV vaccination; HPV&HBV vaccin

SUMMARY:
Rationale:

In march 2009 the Dutch Health Council advised to introduce general infant hepatitis B (HBV) vaccination in the Dutch national immunization program (NIP) {Gezondheidsraad 2009 #16914}. To reach the anticipated health benefits earlier, a catch-up vaccination in pre-adolescents should complement the program, for girls preferably combined with human papillomavirus (HPV) vaccination at the age of 12 years. Although the rationale is clear, particular aspects of combining HPV and HBV vaccination deserve further attention, especially as it has been shown that combining HPV and HBV vaccination results in reduced HBV immunogenicity/seroresponses {Wheeler, Bautista, et al. 2008 #17284}{Pedersen 2009 #16684}. The reason for this interference is unknown, but might be due to concomitant use of different antigens and/or adjuvants, possibly skewing immunity in opposite directions. Despite proven immunostimulatory effects, the use of (new) adjuvants has raised safety concern among the general public as well {Israeli, Agmon-Levin, et al. 2009 #16924}.

Objective, Study design and Study population:

In view of the observations and concerns mentioned above, further investigation into interference of HPV and HBV vaccination and adjuvant use is justified. In this context RIVM propose to study single vs simultaneous HBV and HPV vaccination in 11-12-year-old girls while monitoring antigen-related and antigen-unrelated immunological parameters. The anticipated results will elucidate the extent of interference between simultaneous HPV and HBV vaccination in the target group, and guide the choice for a HBV vaccine and schedule when the HBV catch-up program is indeed introduced. Furthermore, specific immunological trends post single and combined HPV and HBV vaccination will be elucidated, increasing the investigators comprehension of adjuvant use.

ELIGIBILITY:
Inclusion Criteria:

1. Female pre-adolescents born in 1998, eligible for HPV vaccination in 2011.
2. Able to fulfill all study requirements.

Exclusion Criteria:

1. Previous vaccination with any licensed or experimental HPV or HBV vaccine.
2. Contraindication for vaccination with Cervarix®.
3. Contraindication for vaccination with Engerix-B®.
4. Use of investigational vaccine or medication within 30 days before study
5. History of severe adverse reaction associated with a vaccine or vaccine component.
6. Heart disease
7. Liver disease
8. Spleen removal
9. Asthma
10. Immune deficiency or suppression

Ages: 11 Years to 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Antibody seroprotection proportion for HBV in groups 1, 2 and 3 measured in Sample 2. | Month 7